CLINICAL TRIAL: NCT02554032
Title: A Randomized Controlled Trial of Axillary vs. Innominate Artery Cannulation for Antegrade Cerebral Protection in Aortic Surgery: The ACE Randomized Trial
Brief Title: The Aortic Surgery Cerebral Protection Evaluation (ACE) Randomized CardioLink-3 Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-071
Record Dates: First submitted 2015-06-10; First posted 2015-09-18 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Aortic Aneurysm, Thoracic
Keywords: antegrade cerebral perfusion; innominate artery cannulation; axillary artery cannulation; aortic surgery; deep hypothermic circulatory arrest
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Axillary artery cannulation (Active Comparator): Axillary artery cannulation for antegrade cerebral perfusion
  Interventions: Procedure: Axillary artery cannulation
- Innominate artery cannulation (Active Comparator): Innominate artery cannulation for antegrade cerebral perfusion
  Interventions: Procedure: Innominate artery cannulation

INTERVENTIONS:
Procedure: Axillary artery cannulation — The right axillary artery will be exposed via an infraclavicular incision and a Dacron graft sewn to it in an end to side fashion after 5000 units of IV heparin. Following median sternotomy and full systemic heparinization, CPB will be initiated and the patient cooled. The base of the innominate artery will be clamped, and antegrade cerebral perfusion will be provided via the axillary artery. Following completion of the distal open aortic anastomosis, the clamp on the innominate artery will be removed, CPB via the aorta will be resumed and the patient will be rewarmed. After completion of surgery and weaning from CPB, the axillary artery graft will then be removed, the artery repaired and the skin will be closed.
  Arms: Axillary artery cannulation
Procedure: Innominate artery cannulation — After median sternotomy, systemic heparinization, cannulation of the ascending aorta and right atrium, CPB and systemic cooling will be initiated. The ascending aorta, proximal arch and the base of the innominate artery will be mobilized. Purse-string sutures are placed on the anterior wall of the proximal innominate artery and a pediatric venous cannula inserted using a J wire and sequential dilatation. Circulatory arrest with ACP is provided by clamping the base of the innominate artery and connecting the afferent limb of the CPB circuit to the innominate cannula. Once the distal aortic anastomosis is completed, ACP is discontinued, and full CPB via the aortic graft is resumed. Rewarming and the remaining surgery are then completed.
  Arms: Innominate artery cannulation

SUMMARY:
The ACE trial is a multicentre, randomized controlled trial comparing axillary vs. innominate artery cannulation for established antegrade cerebral perfusion in patients having aortic surgery (thoracic and aortic arch) requiring deep hypothermic circulatory arrest using a non-inferiority trial design.

DETAILED DESCRIPTION:
Surgery on the thoracic aorta often requires a brief period of deep hypothermic circulatory arrest (DHCA). The most feared complication of aortic surgery is neurological injury, which can range from mild cognitive impairment to more severe injuries such as stroke. Due to the significant morbidity and mortality associated with post-operative stroke and neurological dysfunction, cerebral protection techniques have evolved extensively. A recommended approach to cerebral protection during DHCA is to deliver blood to the brain in an antegrade fashion via the arterial system, so called antegrade cerebral perfusion (ACP). Axillary artery cannulation, a form of ACP, has become the preferred method of neuroprotection for aortic operations requiring DHCA. However, axillary artery cannulation requires more surgical time and presents potential complications such as brachial plexus injury, seromas, and limb ischemia. The present study aims to determine whether a less common alternative strategy, innominate artery cannulation, offers similar neuroprotection compared to axillary artery cannulation and reduces operative times. A total of 110 patients undergoing elective aortic surgery will be randomly assigned to one of the two strategies. The primary outcome will be the number of patients with new ischemic lesions found on post-operative diffusion weighted MRI (DW-MRI) and total operative time.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Elective aortic arch operation.
3. Planned open distal anastamosis with deep hypothermic circulatory arrest.

Exclusion Criteria:

1. Patients undergoing surgery for aortic dissection or urgent/emergent operation.
2. Patients undergoing surgery for total aortic arch replacement.
3. Patients who are unable to undergo MRI scan (such as due to claustrophobia).
4. Use of an investigational drug or device at the time of enrolment
5. Participation in another clinical trial which interferes with performance of the study procedures or assessment of the outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
new severe ischemic lesions | Post-operative day 4
  The primary safety endpoint of this trial is the proportion of patients with new severe ischemic lesions found on post-operative DW-MRI compared with pre-operative MRI.
Total operative time | Intra-operative
  The primary efficacy endpoint of this trial is the difference in total operative time between the innominate artery cannulation group and the axillary artery cannulation group.

SECONDARY OUTCOMES:
all-cause mortality | 30-day
Stroke or TIA (transient ischemic attack) | 30-day
Neurocognitive dysfunction | Post-operative day 4
  Montreal Cognitive Assessment (MOCA) and Mini-Mental State Examination (MMSE)
Number of new ischemic lesions | Post-operative day 4
  assessed by DW-MRI
Volume of new ischemic lesions | Post-operative day 4
  assessed by DW-MRI
Intracerebral hemorrhage | Post-operative day 4
  assessed by DW-MRI
S100B and Neuron Specific Enolase | 24 hours post-op
  Post-operative serum level of circulating biomarkers of neuronal injury
Post-operative sepsis, delirium, seizure, encephalopathy, atrial fibrillation, post-operative myocardial infarction, re-operation | 30-day
Seroma, brachial plexus injury, reduced arm mobility and pain, arm ischemia | 30-day

OTHER OUTCOMES:
Cerebral oximetry desaturation | intra-operative
CPB (cardiopulmonary bypass) time | intra-operative
Deep hypothermic circulatory arrest time | intra-operative
Antegrade cerebral perfusion time | intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: David Mazer, MD, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - St Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Chen CH, Peterson MD, Mazer CD, Hibino M, Beaudin AE, Chu MWA, Dagenais F, Teoh H, Quan A, Dickson J, Verma S, Smith EE. Acute Infarcts on Brain MRI Following Aortic Arch Repair With Circulatory Arrest: Insights From the ACE CardioLink-3 Randomized Trial. Stroke. 2023 Jan;54(1):67-77. doi: 10.1161/STROKEAHA.122.041612. Epub 2022 Oct 31. PMID 36315249
- [Derived] Peterson MD, Garg V, Mazer CD, Chu MWA, Bozinovski J, Dagenais F, MacArthur RGG, Ouzounian M, Quan A, Juni P, Bhatt DL, Marotta TR, Dickson J, Teoh H, Zuo F, Smith EE, Verma S; ACE CardioLink-3 Trial Working Group. A randomized trial comparing axillary versus innominate artery cannulation for aortic arch surgery. J Thorac Cardiovasc Surg. 2022 Nov;164(5):1426-1438.e2. doi: 10.1016/j.jtcvs.2020.10.152. Epub 2020 Dec 1. PMID 33431219
- [Derived] Garg V, Peterson MD, Chu MW, Ouzounian M, MacArthur RG, Bozinovski J, El-Hamamsy I, Victor Chu F, Garg A, Hall J, Thorpe KE, Dhingra N, Teoh H, Marotta TR, Latter DA, Quan A, Mamdani M, Juni P, David Mazer C, Verma S. Axillary versus innominate artery cannulation for antegrade cerebral perfusion in aortic surgery: design of the Aortic Surgery Cerebral Protection Evaluation (ACE) CardioLink-3 randomised trial. BMJ Open. 2017 Jun 10;7(6):e014491. doi: 10.1136/bmjopen-2016-014491. PMID 28601820